CLINICAL TRIAL: NCT06238440
Title: Comparison of the Efficacy of Different Treatment Approaches in Carpal Tunnel Syndrome: Randomized Controlled Double-Blind Study
Brief Title: Comparison of Different Treatment Approaches in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Banu BAYAR, Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/XIV
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome; Splints; Rigid Taping; Kinesiotape
Keywords: functionality; grip strength; Pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Splints

STUDY DESIGN:
Intervention Model Description: Prospective. A randomized controlled double-blind study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): In the control group (CG), a conventional physiotherapy program will be implemented for 2 weeks. A 10-session treatment will be completed using thermal and electrical agents specified in the program prescribed by the physiotherapist.
  Interventions: Other: Splint and taping methods
- Splint (Experimental): In the Splint (SP) group, in addition to the 10-session conventional physiotherapy program, individuals will be instructed to use the splint prescribed by the physician for 2 weeks.
  Interventions: Other: Splint and taping methods
- Rigid taping (Experimental): In the Rigid taping (RB) group, along with the 10-session conventional physiotherapy program, a rigid strapping application will be performed by an experienced researcher at the end of each physiotherapy session, five days a week.
  Interventions: Other: Splint and taping methods
- Kinesiotape (Experimental): In the Kinesiotape (KT) group, in addition to the 10-session conventional physiotherapy program, kinesiotape application will be carried out by a certified researcher. To ensure homogeneity, individuals in both strapping groups will be asked to remove the tape before coming to treatment and reapply it at the end of the session.
  Interventions: Other: Splint and taping methods

INTERVENTIONS:
Other: Splint and taping methods — In the control group (CG), a conventional physiotherapy program will be implemented for 2 weeks. A 10-session treatment will be completed using thermal and electrical agents specified in the program prescribed by the physiotherapist.
  Splint group: CG + Splint Rigid taping group: CG+ Rigid taping Kinesiotape: CG+ kinesiotape

SUMMARY:
The effectiveness of various external applications (strapping and splinting) on grip strength, pain intensity, symptom level, and functional status in carpal tunnel syndrome (CTS) has been compared in this study. Comparative testing was conducted with exercise and mobilization applications (carpal bone mobilization, yoga, tendon and nerve gliding exercises, neurodynamic mobilization, instrument-assisted soft tissue massage, and standard soft tissue massage) in control groups, placebo groups, and groups undergoing other non-surgical treatments (orthotic application, steroid injections, and other physical agents). Criticisms regarding these studies include bias, lack of blinding, and small intergroup differences. In the literature, evidence supporting the beneficial effects of splinting and strapping applications on CTS is reported to be of low quality, emphasizing the need for higher-quality studies. In light of the information obtained, this study aims to compare the effects of different external applications (strapping and splinting) on grip strength, pain intensity, symptom level, and functional status in CTS.

DETAILED DESCRIPTION:
The inclusion of 40 volunteers is planned for the study. Participants will be divided into four groups, namely control, splint, rigid strapping, and kinesiotape, with the intention of having 10 participants in each group using the closed envelope method.

In the control group (CG), a conventional physiotherapy program will be implemented for 2 weeks. A 10-session treatment will be completed using thermal and electrical agents specified in the program prescribed by the physiotherapist.

In the Splint (SP) group, in addition to the 10-session conventional physiotherapy program, individuals will be instructed to use the splint prescribed by the physician for 2 weeks.

In the Rigid Strapping (RB) group, along with the 10-session conventional physiotherapy program, a rigid strapping application will be performed by an experienced researcher at the end of each physiotherapy session, five days a week.

In the Kinesiotape (KT) group, in addition to the 10-session conventional physiotherapy program, kinesiotape application will be carried out by a certified researcher. To ensure homogeneity, individuals in both strapping groups will be asked to remove the tape before coming to treatment and reapply it at the end of the session. All participants included in the study will be evaluated twice, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* To be volunteered
* To be in the age range of 18-65
* To be diagnosed with mild to moderate carpal tunnel syndrome (CTS) through median nerve conduction velocity studies
* To have experienced paresthesia, pain, and vasomotor symptoms in the area associated with the N. medianus for more than six weeks, as determined by studies on median nerve conduction.
* To test positive in Phalen, Tinel, or carpal compression tests
* To have been recommended splint therapy for CTS

Exclusion Criteria:

* Having a distal motor latency of the median nerve of less than 4.2 milliseconds and/or a distal sensory latency of less than 3.2 milliseconds as a result of electrodiagnostic studies on nerve conduction velocity
* History of malignant tumor
* Use of a pacemaker
* Presence of severe electrodiagnostic findings (fibrotic changes in the median nerve)
* Another inflammatory condition (rheumatoid arthritis, tendinitis, etc.)
* Osteoarthritis in the hand/wrist
* Any musculoskeletal conditions affecting the hand, elbow, or wrist
* Yhyroid dysfunction
* Diagnosis of chronic kidney failure and undergoing treatment for it
* History of carpal tunnel surgery, upper extremity, and neck surgery and trauma
* Diagnosis of carpal tunnel syndrome associated with pregnancy or diabetes
* Having received any treatment for carpal tunnel syndrome (splint therapy, physical agents, exercise, local corticosteroid injection) up to 3 months before the tests
* Hypersensitivity (allergy to Kinesiotape or rigid strapping)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65
Enrollment: 40 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Visuai Analog Scale (VAS) | Baseline- after two weeks
  Pain
Boston Carpal Tunnel Syndrome Questionnaire | Baseline- after two weeks
  Symptom and Function
Handgrip Dynamometer | Baseline- after two weeks
  Grip

CONTACTS AND LOCATIONS:
Overall Officials: Özge ipek Dongaz, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not a study that requires sharing of personal data. Participants' data regarding the study will be given anonymously during publication.